CLINICAL TRIAL: NCT00726934
Title: The Effectiveness of the Neutropenic Diet in Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Karen Moody, Director of Pediatric Palliative Care, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 06-08-367
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Non-Hodgkins Lymphoma; Sarcoma; Neuroblastoma
Keywords: Neutropenic Diet; Food Safety Guidelines; child; cancer
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Sarcoma; Neuroblastoma; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neutropenic Diet (Active Comparator): Participants will be instructed to follow a Neutropenic Diet. This group will receive the same information as the Food Safety Arm with some additional recommendations for avoiding high bacteria foods during length of time on study.
  Interventions: Other: Food Safety Guidelines; Other: Neutropenic Diet
- FDA Food Safety Guidelines (Active Comparator): Participants will be instructed to follow the FDA Food Safety Guidelines
  Interventions: Other: Food Safety Guidelines

INTERVENTIONS:
Other: Food Safety Guidelines — Participants will be randomized to the food safety guidelines will receive information and recommendations regarding Food Shopping, Food Storage, Food Preparation, Safe Cooking, and Safe Serving of Food.
  Other Names: Food Safety Diet; FDA Food Safety Guidelines
Other: Neutropenic Diet — The Neutropenic Diet Guideline includes all information contained in the FDA Food Safety Guidelines with the addition of the following recommendations:
  1. Avoid raw vegetables and fruit (Oranges and bananas are okay.)
  2. Avoid take-out foods and fast foods and fountain drinks.
  3. Avoid aged cheese (blue, Roquefort, Brie).
  4. Cook all produce to well done. Eggs must be hard-boiled.
  5. Avoid deli meats.
  6. No raw nuts, nuts roasted in shell, or freshly ground nut butters from a health food store.
  7. No well water
  8. No yogurt
  Other Names: Low Bacteria Diet
  Arms: Neutropenic Diet

SUMMARY:
The purpose of this study is to determine if FDA approved food safety guidelines are equivalent to a low bacterial diet (the neutropenic diet) with respect to the acquisition of infections during neutropenia in a sample of pediatric cancer patients.

DETAILED DESCRIPTION:
Historically, many interventions have been tried to reduce the incidence of infection by reducing patients' exposures to potential pathogens. The neutropenic diet is one such intervention that was intended to reduce the introduction of bacteria into the host's gastrointestinal tract. This diet excludes foods considered to be high risk for bacterial colonization, especially raw fruits and vegetables. The only studies evaluating this diet have used this intervention in combination with germ free environments, which have been phased out of practice, and the independent effect of this diet remains unknown. In addition, pediatric oncology patients suffer significant gastrointestinal side effects secondary to cancer therapy, which are likely to affect their satisfaction with this dietary regimen. Qualitative data in these children suggests that decreased pleasure from food is a major concern for them and preliminary data on the neutropenic diet showed that although patients were able to stick to it, they found it difficult. The Centers for Disease Control (CDC) and the Food and Drug Administration (FDA) offer more liberalized food safety guidelines for immunocompromised patients. We hypothesize that the neutropenic dietary restrictions offer no advantage over the FDA and CDC endorsed food safety guidelines and that the food safety guidelines will afford patients an improved quality of life through increased choice and control over their diet. The results of this study could potentially modify clinical practice to improve the quality of life of these patients without adverse effects on their rate of infection. Furthermore, the allowance of fresh fruits and vegetables back into the diets of these patients may have a positive impact on their health.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 1 and 30 years with:

   * Acute lymphoblastic leukemia/lymphoma
   * Malignant brain tumor
   * Non-CNS solid tumors
   * Acute myeloblastic leukemia
   * Non-Hodgkin's lymphoma Hodgkin's disease
   * Head and Neck tumors
2. Patients MUST also be ready to receive a cycle of chemotherapy that predictably renders neutropenia at least 70% of the time OR has a risk of febrile neutropenia of at least 20%. This can be any cycle number, it does NOT need to be the FIRST cycle of chemotherapy they are to receive.

Exclusion Criteria:

* Patients receiving myeloablative chemotherapy in preparation for allogeneic or autologous bone marrow or stem cell transplant.
* Co-morbidity with immunosuppressive disease such as AIDS.
* Asplenia.
* Patients with documented infection at time of enrollment.
* Patients who are not fed orally (G-tube dependant, TPN-dependant).
* Patients actively receiving radiation to the brain or gastrointestinal tract for sarcoma.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 2007-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Neutropenic Infection | approximately 4 weeks

SECONDARY OUTCOMES:
Documented Infection | approximately 4 weeks
Quality of life | Baseline and at study end

CONTACTS AND LOCATIONS:
Overall Officials: Karen Moody, MD, MS, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - Rady Children's Hospital San Diego, San Diego, California
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York